CLINICAL TRIAL: NCT05491031
Title: Evaluation of MRI Biomarkers Predictive of Disability Progression in Patients With Multiple Sclerosis
Brief Title: MRI Biomarkers Predictive of Disability Progression in Patients With Multiple Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MR7T-PRADIMS
Record Dates: First submitted 2022-04-05; First posted 2022-08-08 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis; Magnetic Resonance Spectroscopy
Keywords: Multiple sclerosis; ultra-high field 7T magnetic resonance spectroscopy; sodium imaging; predictive MR biomarker of MS
MeSH Terms: conditions — Multiple Sclerosis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multiple sclerosis (Experimental)
  Interventions: Other: magnetic resonance spectroscopy

INTERVENTIONS:
Other: magnetic resonance spectroscopy — Investigation of the association, in patients with multiple sclerosis, between MRI biomarker data at inclusion and progression of physical disability during follow-up (6, 12, 18 and 24 months) assessed by a composite endpoint EDSS plus (EDSS, 9HPT, T25FW)

SUMMARY:
The transition from relapsing-remitting multiple sclerosis to secondarily progressive multiple sclerosis (SPMS) is difficult to identify. Typically, SPMS is diagnosed retrospectively, with a significant delay, on the basis of a clinical history of progressive worsening, independent of relapses. Thus, SPMS is often associated with a considerable period of diagnostic uncertainty.

The use of ultra-high field imaging can shed light on the mechanisms of disability progression thanks to its better spatial resolution and advanced imaging techniques.

The new morphological imaging techniques make it possible to visualize chronic inflammatory lesions and to evaluate their evolution. It also allows for the precise measurement of brain atrophy, a reference in the evaluation of neurodegeneration.

Metabolic imaging via proton spectroscopy allows the analysis of several promising cerebral metabolites that can provide information on cellular energy metabolism, mitochondrial function, or oxidative stress, and can help identify tissues at risk of neurodegeneration. Sodium imaging can provide information on axonal energy metabolism before the occurrence of stable and irreversible axonal damage. This technique is promising as an early marker of neurodegeneration.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* Duration of disease ≤ 25 years,
* Irreversible disability ≤ 7 (permanent wheelchair use) on the EDSS scale

Exclusion Criteria:

* Other progressive neurological disease,
* Isolated radiologic syndrome (RIS),
* Severe psychiatric pathology not in balance,
* Change in dosage, discontinuation or initiation of a psychotropic treatment within the last month,
* Change in background MS treatment for less than 3 months,
* A course of corticosteroids (oral or intravenous) for less than one month,
* Patient with a contraindication to MRI: pregnancy, metallic ocular foreign body (accidental splinters or others), pacemaker, implantable defibrillator, neurostimulator not compatible with MRI 7.0 T, cochlear implants and in general any electronic medical equipment implanted in an irremovable way: metallic cardiac valve, vascular clips (formerly implanted on cranial aneurysm), metallic prosthesis...),
* Illiterate and non-French speaking patient: patient who is partially or completely unable to read and write French.
* Patient benefiting from reinforced protection, i.e. minor, subject deprived of liberty by a judicial or administrative decision, subject staying in a health or social establishment, adult under legal protection and finally patient in emergency situation,
* Pregnant or breastfeeding women, women of childbearing age who do not have effective contraception (hormonal/mechanical: per os, injectable, transcutaneous, implantable, intrauterine device, or surgical: tubal ligation, hysterectomy, total oophorectomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Identify imaging biomarkers at inclusion predictive of disability progression. | up to 24 months
  Determine the correlation between biomarkers concentrations (in mmol/L) with physical disability at inclusion and during follow-up (6, 12, 18 and 24 months) in patients with multiple sclerosis.
  Physical disability is assessed by an Expanded Disability Status Scale plus (EDSS-plus). EDSS-Plus defined as progression on ⩾1 of 3 components (T25FW, 9HPT, EDSS). EDSS score is ordinal rating system ranging from 0 (normal neurological status) to 10 (death), Timed 25-Foot Walk test (T25FW) (second) and 9-Hole Peg Test (9HPT) based on the time for patient to take the 9 pegs and place them in the holes (second).

SECONDARY OUTCOMES:
Determine the correlation between brain MRI and the concentration of imaging biomarkers (mmols) at 6, 12, 18 and 24 months. | up to 24 months
Develop realistic mathematical models of disease progression associated with clinical assessment of disability through dynamics, by the EDSS-plus score (EDSS scale from 0 to 10, T25FW in seconds, 9HPT in seconds). | up to 24 months
  Mathematical models of disease progression using the concentration of biomarkers (in mmol) associated with clinical evaluation of disability (EDSS-plus) over a dynamic period.
Develop an artificial intelligence algorithm to identify predictive markers for disability. The artificial intelligence algorithm utilizes patients' clinical (EDSSS-Plus Scale) and radiological (brain MRI) characteristics. | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- PoitiersUH, Poitiers, France